CLINICAL TRIAL: NCT03426384
Title: Can Individualized Diet and Lifestyle Modifications Derived From Digital Therapeutics and Health Coaching Improve Symptoms of Systemic Lupus Erythematosus
Brief Title: FLARE Lupus Research Study Systemic Lupus Erythematosus
Acronym: FLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mymee Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20172250
Record Dates: First submitted 2018-01-18; First posted 2018-02-08 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: System; Lupus Erythematosus
Keywords: SLE; FLARE; Lupus; Digital Therapeutics; Health Coaching; Smartphone App
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The Intervention Group will enter daily tasks into the Mymee app. After the first intake session, the subject will participate in weekly 20-30-minute coaching sessions with the Health Coach. At the second session, the Health Coach will review the symptoms and the free text entered by the subject to determine which dietary and environmental factors will be monitored in the Mymee app.
  Each subsequent week, the Health Coach will review and discuss with the subject the food diary and the data entered into the Mymee app during the previous week. Based on this discussion and the subject's medical records, the Health Coach will determine or revise which symptoms will continue to be monitored using the Mymee App.
  Interventions: Behavioral: Mymee Program
- Control Group (No Intervention): The Control Group subjects will receive no training, coaching, or other intervention services from Mymee. The Control Group subjects will complete the same battery of assessments at the same intervals as the Intervention Group subjects.

INTERVENTIONS:
Behavioral: Mymee Program — A combination of digital therapeutics and telephonic health coaching is used to identify and test dietary, lifestyle, and environmental triggers in order to reduce symptoms of auto-immune disease.
  Arms: Intervention Group

SUMMARY:
The first phase of this pilot study will assess changes in quality of life at the end of a 16-week Mymee program in patients with moderate to severe SLE. The second phase will assess changes in healthcare utilization and cost over a one year period after program end.

DETAILED DESCRIPTION:
Intervention Group The Intervention Group will enter daily tasks into the Mymee app. After the first intake session, the subject will participate in weekly 20-30-minute coaching sessions with the Health Coach. At the second session, the Health Coach will review the symptoms and the free text entered by the subject to determine which dietary and environmental factors will be monitored in the Mymee app.

Each subsequent week, the Health Coach will review and discuss with the subject the food diary and the data entered into the Mymee app during the previous week. Based on this discussion and the subject's medical records, the Health Coach will determine or revise which symptoms will continue to be monitored using the Mymee App.

Control Group The Control Group subjects will receive no training, coaching, or other intervention services from Mymee. The Control Group subjects will complete the same battery of assessments at the same intervals as the Intervention Group subjects.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age who can consent for themselves
* Location - U.S.
* Proficient in English (speaking, reading, and writing)
* Own or have reliable access to a smartphone (iPhone or Android)
* Provision of medical record
* Diagnosis of Lupus SLE as indicated in medical record
* Symptomatic lupus as indicated by a score of at least 6 on one or more of BPI-SF questions 3, 5, or 6 and/or a score of at least 3 on one or more of the first four questions on the FACIT
* Current prescription for one or more of the following medications: 20mg/day of oral prednisone (or other oral corticosteroid equivalent dose); methotrexate and/or other immunosuppressive therapy of any dosage such as cyclophosphamide (Cytoxan®), methotrexate (Rheumatrex™), or azathioprine (muran®), adalimumab (Humira Pen, Humira Pen Crohn's-UC-HS Start, Humira Pediatric Crohn's Start, Humira, and Humira Pen Psoriasis-Uveitis), Plaquenil, Cellcept; monoclonal antibodies (mAbs) such as Benlysta® (belimuab, formerly called LymphoStat-B™); rituximab (Rituxan, MabThera and others);
* Able and willing to consent to study protocol
* Medications which have been stable for 3 months

Exclusion Criteria:

* Pregnant and/or planning to get pregnant before end of 16-week intervention
* In prison during any part of the 16-month study period
* Resident of a nursing home, wards of the state, or Institutionalized during any part of the 16-month study period
* Persons with decisional incapacity/cognitive impairment
* Participating in another clinical trial, interventional or observational research during the study period
* Plan or intention to receive/start during the 16-week (112 day) intervention period either:

  1. a standing dose of oral steroid agents at a 20mg dose of prednisone (or other oral corticosteroid equivalent dose);
  2. pulses or tapers of steroids for flares for more than a total of 30 days within the observation period
  3. any pulse/taper dose of steroids during the last 4 weeks of the intervention period;
  4. immunosuppressive agents, or biologic response modifiers.
* Diagnosed with cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form (BPI-SF) | Change from baseline, measured at weeks 4, 8, 12, and 16 of the intervention and then every 3 months for the 1 year following the intervention
  BPI-SF is a 9-item questionnaire with two domains: pain severity and pain interference. The pain severity items have values which range from 0 ("no pain") to 10 ("pain as bad as you can imagine"), and the pain interference items have values which range from 0 ("does not interfere") to 10 ("completely interferes"). The pain severity and pain interference domain scores can be calculated as the mean of the scores of their component items.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Change from baseline, measured at weeks 4, 8, 12, and 16 of the intervention and then every 3 months for the 1 year following the intervention]
  The FACIT-Fatigue Sale is a 13-item questionnaire assessing fatigue, where the items use a Likert-type scale (with values ranging from 0 to 4). The responses for each item are added to obtain a total score which ranges from 0 to 52, with a higher score indicating less fatigue.
LupusQOL | Change from baseline, measured at weeks 4, 8, 12, and 16 of the intervention and then every 3 months for the 1 year following the intervention
  LupusQoL is a Systemic Lupus Erythematosus (SLE) specific health-related quality of life measure. It is a 34-item questionnaire where each item uses a 5-point Likert-type scale (with values ranging from 0 to 4). Each item pertains to one of eight domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue. Each domain of the LupusQoL is scored separately. The score for each domain is equal to the average of the domain's items scaled such that the range of possible scores is 0 (worst health-related quality of life) to 100 (best health-related quality of life).

SECONDARY OUTCOMES:
Change in healthcare cost | 1 year
  Comparison of healthcare costs over a one year period, pre- and post- intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mymee Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaul A, Gordon C, Crow MK, Touma Z, Urowitz MB, van Vollenhoven R, Ruiz-Irastorza G, Hughes G. Systemic lupus erythematosus. Nat Rev Dis Primers. 2016 Jun 16;2:16039. doi: 10.1038/nrdp.2016.39. PMID 27306639
- [Background] Lim SS, Bayakly AR, Helmick CG, Gordon C, Easley KA, Drenkard C. The incidence and prevalence of systemic lupus erythematosus, 2002-2004: The Georgia Lupus Registry. Arthritis Rheumatol. 2014 Feb;66(2):357-68. doi: 10.1002/art.38239. PMID 24504808
- [Background] Lisnevskaia L, Murphy G, Isenberg D. Systemic lupus erythematosus. Lancet. 2014 Nov 22;384(9957):1878-1888. doi: 10.1016/S0140-6736(14)60128-8. Epub 2014 May 31. PMID 24881804
- [Background] Somers EC, Marder W, Cagnoli P, Lewis EE, DeGuire P, Gordon C, Helmick CG, Wang L, Wing JJ, Dhar JP, Leisen J, Shaltis D, McCune WJ. Population-based incidence and prevalence of systemic lupus erythematosus: the Michigan Lupus Epidemiology and Surveillance program. Arthritis Rheumatol. 2014 Feb;66(2):369-78. doi: 10.1002/art.38238. PMID 24504809
- [Background] Davis LS, Reimold AM. Research and therapeutics-traditional and emerging therapies in systemic lupus erythematosus. Rheumatology (Oxford). 2017 Apr 1;56(suppl_1):i100-i113. doi: 10.1093/rheumatology/kew417. PMID 28375452
- [Background] Pons-Estel GJ, Alarcon GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010 Feb;39(4):257-68. doi: 10.1016/j.semarthrit.2008.10.007. Epub 2009 Jan 10. PMID 19136143
- [Background] Bernatsky S, Boivin JF, Joseph L, Manzi S, Ginzler E, Gladman DD, Urowitz M, Fortin PR, Petri M, Barr S, Gordon C, Bae SC, Isenberg D, Zoma A, Aranow C, Dooley MA, Nived O, Sturfelt G, Steinsson K, Alarcon G, Senecal JL, Zummer M, Hanly J, Ensworth S, Pope J, Edworthy S, Rahman A, Sibley J, El-Gabalawy H, McCarthy T, St Pierre Y, Clarke A, Ramsey-Goldman R. Mortality in systemic lupus erythematosus. Arthritis Rheum. 2006 Aug;54(8):2550-7. doi: 10.1002/art.21955. PMID 16868977
- [Background] Lightstone L, Doria A, Wilson H, Ward FL, Larosa M, Bargman JM. Can we manage lupus nephritis without chronic corticosteroids administration? Autoimmun Rev. 2018 Jan;17(1):4-10. doi: 10.1016/j.autrev.2017.11.002. Epub 2017 Nov 3. PMID 29108828
- [Background] Wild CP. Complementing the genome with an "exposome": the outstanding challenge of environmental exposure measurement in molecular epidemiology. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1847-50. doi: 10.1158/1055-9965.EPI-05-0456. No abstract available. PMID 16103423
- [Background] Squance ML, Reeves GE, Bridgman H. The Lived Experience of Lupus Flares: Features, Triggers, and Management in an Australian Female Cohort. Int J Chronic Dis. 2014;2014:816729. doi: 10.1155/2014/816729. Epub 2014 Nov 20. PMID 26464865
- [Background] Kamen DL. Environmental influences on systemic lupus erythematosus expression. Rheum Dis Clin North Am. 2014 Aug;40(3):401-12, vii. doi: 10.1016/j.rdc.2014.05.003. PMID 25034153
- [Background] Gulati G, Brunner HI. Environmental triggers in systemic lupus erythematosus. Semin Arthritis Rheum. 2018 Apr;47(5):710-717. doi: 10.1016/j.semarthrit.2017.10.001. Epub 2017 Oct 5. PMID 29169635
- [Background] Mu Q, Zhang H, Luo XM. SLE: Another Autoimmune Disorder Influenced by Microbes and Diet? Front Immunol. 2015 Nov 30;6:608. doi: 10.3389/fimmu.2015.00608. eCollection 2015. PMID 26648937
- [Background] Bates MA, Brandenberger C, Langohr II, Kumagai K, Lock AL, Harkema JR, Holian A, Pestka JJ. Silica-Triggered Autoimmunity in Lupus-Prone Mice Blocked by Docosahexaenoic Acid Consumption. PLoS One. 2016 Aug 11;11(8):e0160622. doi: 10.1371/journal.pone.0160622. eCollection 2016. PMID 27513935
- [Background] He B, Hoang TK, Wang T, Ferris M, Taylor CM, Tian X, Luo M, Tran DQ, Zhou J, Tatevian N, Luo F, Molina JG, Blackburn MR, Gomez TH, Roos S, Rhoads JM, Liu Y. Resetting microbiota by Lactobacillus reuteri inhibits T reg deficiency-induced autoimmunity via adenosine A2A receptors. J Exp Med. 2017 Jan;214(1):107-123. doi: 10.1084/jem.20160961. Epub 2016 Dec 19. PMID 27994068
- [Background] Sepah SC, Jiang L, Peters AL. Long-term outcomes of a Web-based diabetes prevention program: 2-year results of a single-arm longitudinal study. J Med Internet Res. 2015 Apr 10;17(4):e92. doi: 10.2196/jmir.4052. PMID 25863515
- [Background] Hsu WC, Lau KH, Huang R, Ghiloni S, Le H, Gilroy S, Abrahamson M, Moore J. Utilization of a Cloud-Based Diabetes Management Program for Insulin Initiation and Titration Enables Collaborative Decision Making Between Healthcare Providers and Patients. Diabetes Technol Ther. 2016 Feb;18(2):59-67. doi: 10.1089/dia.2015.0160. Epub 2015 Dec 8. PMID 26645932
- [Background] McKenzie AL, Hallberg SJ, Creighton BC, Volk BM, Link TM, Abner MK, Glon RM, McCarter JP, Volek JS, Phinney SD. A Novel Intervention Including Individualized Nutritional Recommendations Reduces Hemoglobin A1c Level, Medication Use, and Weight in Type 2 Diabetes. JMIR Diabetes. 2017 Mar 7;2(1):e5. doi: 10.2196/diabetes.6981. PMID 30291062
- [Background] Holloway L, Humphrey L, Heron L, Pilling C, Kitchen H, Hojbjerre L, Strandberg-Larsen M, Hansen BB. Patient-reported outcome measures for systemic lupus erythematosus clinical trials: a review of content validity, face validity and psychometric performance. Health Qual Life Outcomes. 2014 Jul 22;12:116. doi: 10.1186/s12955-014-0116-1. PMID 25048687
- [Background] McElhone K, Abbott J, Sutton C, Mullen M, Lanyon P, Rahman A, Yee CS, Akil M, Bruce IN, Ahmad Y, Gordon C, Teh LS. Sensitivity to Change and Minimal Important Differences of the LupusQoL in Patients With Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2016 Oct;68(10):1505-13. doi: 10.1002/acr.22850. Epub 2016 Sep 2. PMID 26816223
- [Derived] Khan F, Granville N, Malkani R, Chathampally Y. Health-Related Quality of Life Improvements in Systemic Lupus Erythematosus Derived from a Digital Therapeutic Plus Tele-Health Coaching Intervention: Randomized Controlled Pilot Trial. J Med Internet Res. 2020 Oct 20;22(10):e23868. doi: 10.2196/23868. PMID 33079070